CLINICAL TRIAL: NCT05451979
Title: High Intensity Interval Training in Pediatric Heart Transplant Recipients: Evaluating a Novel Telemedicine Video Game-Linked Exercise Platform (MedBIKE™)
Brief Title: HIIT in Pediatric Heart Transplant Recipients (MedBIKE™)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute, Canada (Other); Canadian Donation and Transplantation Research Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00109855
Record Dates: First submitted 2021-11-08; First posted 2022-07-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pediatric ALL; Transplant; Failure, Heart
Keywords: Cardiac rehabilitation; High Intensity Interval Training; Telemedicine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Randomized crossover study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MedBIKE HIIT (Experimental): Participants will complete the baseline assessments and begin the MedBIKE HIIT Exercise Program intervention within 2-weeks. After the completion of the 12-week program, participants will return for follow-up assessments which will be repeated at 6- and 12-months post intervention.
  Interventions: Device: MedBIKE HIIT
- Standard of Care (No Intervention): Participants will complete the baseline assessments and continue with standard of care (no intervention) for 12-weeks then return for a repeat assessment. Participants will then crossover into the MedBIKE HIIT Exercise Program intervention group for 12-weeks. A post-intervention assessment will be completed and follow-up assessments at 6- and 12-months post intervention.

INTERVENTIONS:
Device: MedBIKE HIIT — Participants will complete a high intensity interval training exercise program 3 times a week for 12 weeks (36 sessions total)
  Arms: MedBIKE HIIT

SUMMARY:
Heart transplantation is the long-term treatment for children and adults with advanced heart failure. Post-transplant outcomes have improved over time, such that 50% of pediatric heart transplant recipients (HTR) remain alive with a need for re-transplantation 17-years following the initial transplant. With improved short- and medium-term outcomes, focus has shifted towards optimizing long-term survival and reducing transplant-associated morbidities. This includes strategies aimed at optimizing cardiorespiratory fitness and physical activity levels.

Pediatric and adult HTRs have reduced exercise capacity compared with the general population. Previous groups have shown gradual improvements in heart rate response to exercise and exercise capacity in pediatric HTRs. However, after an initial improvement, exercise capacity appears to plateau, or even decline in pediatric HTRs, and remains sub-optimal compared with the general population.

Most exercise interventions in HTRs to date have focused on moderate-intensity continuous exercise (MICE), with some resistance components incorporated. More recently, high-intensity interval training (HIIT), consisting of short, intense bursts of exercise with rest periods, has been explored in the adult HTR population, with findings to date suggesting that it may yield greater improvements in cardiorespiratory fitness compared with MICE. Exercise interventions, particularly HIIT interventions, have consistently shown clinically important improvements in exercise capacity in adult HTRs that are linked with improved long-term post-transplant outcomes and well-being. Unfortunately, trials of exercise interventions in pediatric HTRs remain lacking. This study team is proposing an assessment of the feasibility of a home-based HIIT exercise program using a novel telemedicine-enable video game linked customizable cycle ergometer (MedBIKE™).

DETAILED DESCRIPTION:
Purpose: To determine the feasibility of MedBIKE™ in a 12-week home-based high intensity interval training program in pediatric heart transplant recipients (HTRs).

Hypothesis: The MedBIKE™ intervention will be feasible, with adequate enrolment of eligible participants (>60%), high session compliance (>80%), and low-drop out rate (~10%), with no adverse events directly related to the intervention. The investigators further hypothesize that the MedBIKE™ HIIT intervention will result in immediate and sustained improvements in exercise capacity, physical activity, self-efficacy towards physical activity, and HRQoL.

Justification: Clinical trials of exercise interventions in pediatric HTRs remains significantly lacking. This lack of literature to date has been identified as a significant knowledge gap in the Canadian Society of Transplantation/CAN-RESTORE recent joint statement. While the findings to date indicate that exercise interventions in pediatric HTRs may show improvements in exercise capacity, numerous knowledge gaps remain. For example, despite promising findings in adult HTRs, HIIT has not yet been studied in pediatric HTRs. Moreover, the effect of exercise interventions on physical activity, HRQoL, and self-efficacy towards physical activity have not been well studied. It is important to evaluate whether a supervised exercise intervention at near-maximal intensity can promote improvements in physical activity self-efficacy that may in turn yield sustained improvements in physical activity. One of the limiting factors for regular participation in post-transplant exercise programs is the necessary time commitment that is intensified in a program with demographics such as ours in Western Canada with many post-transplant children living far from the transplant center and with limited access to exercise facilities. A supervised home-based training program could optimize the time-efficiency and accommodate the patient's routine schedules. Thus, the investigators are proposing an assessment of the feasibility of a home-based HIIT exercise program using a novel telemedicine-enabled video game-linked customizable cycle ergometer (MedBIKE™).

Objectives: (Primary) Evaluate the feasibility of a 12-week, home-based HIIT MedBIKE™ intervention in pediatric HTRs. (Secondary) Evaluate the impact of the MedBIKE™ HIIT intervention on 1) exercise capacity; 2) physical activity; 3) self-efficacy towards physical activity; 4) HRQoL and 5) sustained changes in all secondary outcomes at 6- and 12-months post-intervention.

Research Method: Single-center, randomized crossover feasibility trial with a multi-method approach. Potential participants and families will be approached first by a clinical team member. Participants and parents expressing interest will meet with a research coordinator who, along with one of the investigators and the clinical team will screen for eligibility. Written consent and assent (if applicable) will be obtained from participants who are deemed eligible.

Following recruitment, participants will be administered the PedsQL and CSAPPA questionnaires, an accelerometer will be provided for seven days, and a baseline CPET will be performed or scheduled to occur following completion of the accelerometer assessment. Participants will then be randomized via a 1:1 allocation ratio with permuted blocks of randomly varied sizes either to the immediate MedBIKE™ arm or the immediate control arm (usual care) for 12-weeks, followed by a repeat assessment. Participants in the control arm will then cross-over and complete the 12-week MedBIKE™ HIIT program, followed by a repeat assessment at the completion of the intervention. All post-intervention assessments will occur 3-7 days post-MedBIKE™ intervention (to allow adequate recovery) and accelerometers will be programmed to commence counts 24 hours post-assessment to avoid bias from fatigue from the CPET. Participants will then return for final assessments at 6- and 12-months post-MedBIKE™ intervention. Whenever possible, follow-up assessments will be coordinated with clinical appointments (pediatric HTRs are typically clinically assessed every 3-4 months or more frequently).

The MedBIKE™ program is a first-person interactive videogame in which the participant is 'biking' around a safari collecting animals and will enter a wormhole when completing the high-intensity exercise portion. The participant and clinician applications are Windows WPF applications that run on windows 10 PCs. The participant application also includes a companion app that runs on an Android table. The MedBIKE™ service application is a platform-independent Python application that is run on a a secure Ubuntu Linux instance operated by the University of Alberta's Faculty of Medicine and Dentistry IT department.

A follow-up assessment, identical to that of the baseline (questionnaires, CPET, interviews and a 7-day week wear of an accelerometer) will occur 3-14 days post-intervention. These assessments will be repeated at 6- and 12-months post-intervention.

Plan for Data Analysis: The WHCRI biostatistics group will provide statistical and data analysis support. Continuous data will be summarized as median with first and third quartiles and changes in pre- and post-intervention measures will be evaluated using the Mann-Whitney test. Categorical data will be presented by absolute and relative frequencies (n and %). All statistical analyses will be performed by SAS 9.4 or later (SAS Institute Inc., Cary, NC, USA).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric heart transplant recipients, at least 6-months post heart transplantation
* Aged 10-18 years

Exclusion Criteria:

* Non-English speaking (thus limiting communication during the MedBIKE™ sessions)
* Home environment cannot accommodate the MedBIKE™ system (for example, space limitations)
* History of multiorgan transplant
* Adult unavailable to supervise the home-based exercise sessions
* Episode of clinical antibody- or cellular-mediated rejection within 3-months of the baseline assessment
* Previous involvement in a cardiac rehabilitation or exercise intervention program
* Primary cardiologist has exercise restricted the participant or counsels against participation
* Previous exercise stress test demonstrating sustained arrhythmias, ST segment elevation or depression greater than 3mm, an inappropriate rise in blood pressure (BP) (<20 mmHg) or a systolic BP >200 mmHg, or symptoms of chest pain or syncope
* Resting arterial saturation <85% or oxygen requirements
* Moderate ventricular systolic dysfunction (or worse) at the most recent echocardiogram
* History of chest pain on exertion
* Unrepaired/unpalliated CHD
* Arrhythmias in the last year (including supraventricular tachycardia, ventricular tachycardia, atrioventricular block (Mobitz II or worse))
* New York Heart Association class II or worse symptoms
* Active medical inter-current illness limiting ability to participate
* Cognitive impairment limiting the communication needed for the HIIT program
* Extracardiac or congenital abnormality limiting the participant's functional ability to exercise

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of a 12-week, home-based HIIT MedBIKE™ intervention in pediatric heart transplant recipients. | 12 weeks
  Pediatric heart transplant participants will be provided with a MedBIKE™ system to complete a video game linked 12-week high intensity interval training program equipped with telemedicine capabilities. Feasibility will be defined as adequate recruitment of eligible participants (greater than 60 percent), high session compliance (greater than 80 percent), low drop-out rate (less than 10 percent) and safety in terms of no severe adverse events related to the intervention.

SECONDARY OUTCOMES:
Exercise capacity through the change in VO2peak (mL/kg/min) measured using CPET testing. | 13 months
  CPET (Exercise Stress Test with Spirometry) will be done to measure the VO2peak (mL/kg/min) output of participants. A comparison will be done pre- and post-MedBIKE intervention, as well as 6 and 12-months post, to determine the change in overall VO2peak of participants.
Changes in physical activity, defined as time spent in moderate to vigorous physical activity (MVPA) and sedentary time, measured by wearing an accelerometer for 7-days prior and 7-days post MedBIKE intervention | 13 months
  Participants will be provided with an accelerometer to wear for 7-days prior to the start of the MedBIKE intervention program and again for 7-days post intervention and again at 6 and 12-months post intervention. The accelerometer will measure the time spent in moderate to vigorous physical activity (MVPA) and the sedentary time. A comparison will be done pre- and post-MedBIKE intervention to determine changes in the physical activity levels. The 6-month and 12-month time points will be used for a comparison on the sustained changes of the intervention.
Changes in cardiac specific health-related quality of life will be measured using the PedsQL Cardiac Module questionnaire. | 13 months
  Participants will be asked to complete the PedsQL Cardiac Module questionnaire. This questionnaire is a validated multidimensional instrument to assess cardiac specific health-related quality of life in youth. This questionnaire is scored on a scale of 0-100, where a higher score indicates a better quality of life. These scores will be compared pre- and post-MedBIKE intervention to determine changes in health-related quality of life. The 6-month and 12-month time points will be used for a comparison on the sustained changes of the intervention.
Changes in self efficacy towards physical activity measured on the Children's Self-Perceptions of Adequacy in and Predilection for Physical Activity (CSAPPA) scale. | 13 months
  Participants will be asked to complete the Children's Self-Perceptions of Adequacy in and Predilection for Physical Activity (CSAPPA) scale. This questionnaire consists of 19 questions and is a validated tool designed to assess self-perceptions of adequacy and predilection towards physical activity in youth on a scale of low, moderate and high in terms of attitudes towards physical activity. The overall score of this questionnaire will be compared pre- and post-MedBIKE intervention and again at 6 and 12-months post-intervention to evaluate sustained changes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Khoury, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. All data will be de-identified prior to analysis and publication.

REFERENCES:
- [Result] Khoury M, Phillips DB, Wood PW, Mott WR, Stickland MK, Boulanger P, Rempel GR, Conway J, Mackie AS, Khoo NS. Cardiac rehabilitation in the paediatric Fontan population: development of a home-based high-intensity interval training programme. Cardiol Young. 2020 Oct;30(10):1409-1416. doi: 10.1017/S1047951120002097. Epub 2020 Jul 27. PMID 32716280
- [Derived] Nytroen K, Rolid K. A Review of High-Intensity Interval Training in Heart Transplant Recipients: Current Knowledge and Future Perspectives. J Cardiopulm Rehabil Prev. 2024 May 1;44(3):150-156. doi: 10.1097/HCR.0000000000000847. Epub 2024 Mar 15. PMID 38488139